CLINICAL TRIAL: NCT00165997
Title: The Effects of Radiofrequency Ablation Procedures on Quality of Life in the Pediatric Cohort
Brief Title: Quality of Life in Patients Post Radiofrequency Ablation
Status: Terminated | Type: Observational
Why Stopped: sufficient data collected for significant conclusive results
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Margaret Strieper, Principal Investigator, Emory University
Other Study IDs: 0147-2004
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Radiofrequency Catheter Ablation; Quality of Life; Arrhythmia
Keywords: pediatrics; cardiology; Radiofrequency ablation; structurally normal heart
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Radiofrequency ablation is a procedure done in the Catheterization Laboratory to help correct specific problems that cause the heart to beat faster than it should. Quality of life includes the physical as well as the emotional aspects of a patient. Doctors have always tried to take care of a medical problem with minimal physical and emotional risk. It is assumed that once the medical problem is fixed, the patient will have an improved quality of life. To know if this assumption is true, the investigators are asking children scheduled for this procedure, along with their family, to answer questions before the ablation, then answer the same questions 5-6 months after the ablation.

DETAILED DESCRIPTION:
When a patient (age 5-18 years) is scheduled for an ablation at Children's Healthcare of Atlanta, the research coordinator contacts the family prior to the procedure and describes the study to them, details the goals, benefits versus risks, and answers any questions they may have. Written consent is obtained from the parents. Assent is obtained from the child. Both the parent and child are given the age appropriate Peds QL (tm) Pediatric Quality of Life Inventory, version 4.0. The forms are returned to the research coordinator. If the child is ablated, then 5-6 months after the ablation, the same questionnaire is sent to the child and parent. Data are entered into a database.

ELIGIBILITY:
Inclusion Criteria:

* 5-18 years of age
* English is the primary language
* Scheduled for an ablation at Children's Healthcare of Atlanta
* Normally structured heart

Exclusion Criteria:

* Congenital heart defect
* English is not the primary language
* Children with significant neurocognitive deficits as determined by the investigator

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-02; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret J Strieper, DO, Principal Investigator — Emory University and Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States